CLINICAL TRIAL: NCT03437785
Title: A Phase 2, Multi-center, Randomized, Double-blind, Parallel-group Trial to Evaluate the Efficacy and Safety of CKD-495 in Patients With Acute and Chronic Gastritis
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of CKD-495 Tablet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 174AG/CG17002
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-02

CONDITIONS: Gastritis
Keywords: Acute Gastritis; Chronic Gastritis; Cinnamic acid; CKD-495
MeSH Terms: conditions — Gastritis | interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Group 1 (Experimental): Patients assigned to this group are treated with CKD-495 75mg Tab.,and other 3 Placebo Tab.(Placebo of the CKD-495 150mg, ,Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg Tab., Placebo of the Rebamipide 100mg Tab.)
  Interventions: Drug: CKD-495 75mg; Drug: Placebo of the CKD-495 150mg; Drug: Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg; Drug: Placebo of the Rebamipide 100mg
- Experimental Group 2 (Experimental): Patients assigned to this group are treated with CKD-495 150mg Tab.,and other 3 Placebo Tab.(Placebo of the CKD-495 75mg, Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg Tab., Placebo of the Rebamipide 100mg Tab.)
  Interventions: Drug: CKD-495 150mg; Drug: Placebo of the CKD-495 75mg; Drug: Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg; Drug: Placebo of the Rebamipide 100mg
- Placebo Group (Placebo Comparator): Patients assigned to this group are treated with 4 Placebo Tab.(Placebo of the CKD-495 75mg, Placebo of the CKD-495 150mg, Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg Tab., Placebo of the Rebamipide 100mg Tab.)
  Interventions: Drug: Placebo of the CKD-495 75mg; Drug: Placebo of the CKD-495 150mg; Drug: Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg; Drug: Placebo of the Rebamipide 100mg
- Active comparator Group 1 (Active Comparator): Patients assigned to this group are treated with Artemisiae argyi folium 95% ethanol ext.(20→1) 60mg Tab, and other 3 Placebo Tab.(Placebo of the CKD-495 75mg, Placebo of the CKD-495 150mg, Placebo of the Rebamipide 100mg Tab.)
  Interventions: Drug: Artemisiae argyi folium 95% ethanol ext.(20→1) 60mg; Drug: Placebo of the CKD-495 75mg; Drug: Placebo of the CKD-495 150mg; Drug: Placebo of the Rebamipide 100mg
- Active comparator Group 2 (Active Comparator): Patients assigned to this group are treated with Rebamipide 100mg Tab.,and other 3 Placebo Tab.(Placebo of the CKD-495 75mg, Placebo of the CKD-495 150mg, Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg Tab.)
  Interventions: Drug: Rebamipide 100mg; Drug: Placebo of the CKD-495 75mg; Drug: Placebo of the CKD-495 150mg; Drug: Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg

INTERVENTIONS:
Drug: CKD-495 75mg — CKD-495 75mg Tab.
  Arms: Experimental Group 1
Drug: CKD-495 150mg — CKD-495 150mg Tab.
  Arms: Experimental Group 2
Drug: Artemisiae argyi folium 95% ethanol ext.(20→1) 60mg — Artemisiae argyi folium 95% ethanol ext.(20→1) 60mg Tab.
  Arms: Active comparator Group 1
Drug: Rebamipide 100mg — Rebamipide 100mg Tab.
  Arms: Active comparator Group 2
Drug: Placebo of the CKD-495 75mg — Placebo of the CKD-495 75mg Tab.
  Arms: Active comparator Group 1; Active comparator Group 2; Experimental Group 2; Placebo Group
Drug: Placebo of the CKD-495 150mg — Placebo of the CKD-495 150mg Tab.
  Arms: Active comparator Group 1; Active comparator Group 2; Experimental Group 1; Placebo Group
Drug: Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg — Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg Tab.
  Arms: Active comparator Group 2; Experimental Group 1; Experimental Group 2; Placebo Group
Drug: Placebo of the Rebamipide 100mg — Placebo of the Rebamipide 100mg Tab
  Arms: Active comparator Group 1; Experimental Group 1; Experimental Group 2; Placebo Group

SUMMARY:
To Evaluate the Efficacy and Safety of CKD-495

DETAILED DESCRIPTION:
A Phase 2, Multi-center, Randomized, Double-blind, Parallel-group Trial to Evaluate the Efficacy and Safety of CKD-495 in Patients with Acute and Chronic Gastritis

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects aged ≥ 19
2. Acute or Chronic gastritis patients who have more than 1 erosion on endoscopy within 7days prior to the use of the Investigator's Product taken date
3. Patients who have more than 1 subjective symptom

Exclusion Criteria:

1. Patients with peptic ulcer, gastroesophageal reflux disease, malignant tumor in the digestive system or coagulation disorder, or taking antithrombotic medicine
2. Patients who have been taken any gastritis medicine that could affect the treatment: H2 receptor antagonist, PPI(Proton Pump Inhibitor), antacid, improvement of movement in digestive system, Prostaglandin, and protective agent for gastritis
3. Patients who have to take medicine that could cause gastritis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Improvement rate of gastric erosion | 14days after drug administrations
  50% decreased on erosive grade

SECONDARY OUTCOMES:
cure rate of gastric erosion | 14days after drug administrations
  0 erosion
Improvement rate of symptoms | 14days after drug administrations
  50% decreased on the Subjective Symptoms total score
Improvement rate of gastric edema | 14days after drug administrations
  50% decreased on the Edema grade
Improvement rate of gastric erythema | 14days after drug administrations
  50% decreased on the Erythema grade
Improvement rate of gastric hemorrhage | 14days after drug administrations
  50% decreased on the Hemorrhage grade

CONTACTS AND LOCATIONS:
Locations (16):
- South Korea (16):
  - Chonnam National University Hospital, Gwangju, Donggu, Jebongro
  - Keimyung University Dongsan Medical Center, Daegu, Gyeongsangbuk-do
  - Kyungpook National University Hospital, Daegu, Gyeongsangbuk-do
  - Kosin University Gospel Hospital, Busan, Seo-gu
  - Busan National University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Hallym University Chuncheon Seonsim Hospital, Chuncheon
  - Yeungnam University Medical Center, Daegu
  - Wonkwang University Hospital, Iksan
  - Jeju National University Hospital, Jeju City
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Hanyang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SH, Lee OY, Lee YC, Park KS, Park JJ, Park MI, Song GA, Lee DH, Jung H, Kim SK, Kim TN, Choi SC, Jee SR, Rew JS, Lee ST, Choi EK, Baik GH, Park SJ. A Phase 2, Multi-Center, Randomized, Double-Blind, Parallel-Group Trial to Evaluate the Efficacy and Safety of CKD-495 in Patients With Acute and Chronic Gastritis. Can J Gastroenterol Hepatol. 2025 Apr 10;2025:2702089. doi: 10.1155/cjgh/2702089. eCollection 2025. PMID 40255536